CLINICAL TRIAL: NCT03222843
Title: A Phase III,Multicentre, Randomized, Double-Blind and Open-Label Study to Evaluate the Safety and Efficacy of Hetrombopag Olamine in Patients With Idiopathic Thrombocytopenic Purpura
Brief Title: Multicentre, Randomised Phase III Study of the Efficacy and Safety of Hetrombopag Olamine in Idiopathic Thrombocytopenic Purpura (ITP) Patient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-TPO-III-ITP
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2017-07

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): oral hetrombopag at an initial dose of 2.5 mg once daily
  Interventions: Drug: Hetrombopag Olamine
- Arm 2 (Experimental): oral hetrombopag at an initial dose of 5 mg once daily
  Interventions: Drug: Hetrombopag Olamine
- Arm 3 (Placebo Comparator): oral placebo at an initial dose of 2.5 mg once daily
  Interventions: Drug: matching placebo
- Arm 4 (Placebo Comparator): oral placebo at an initial dose of 5 mg once daily
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: Hetrombopag Olamine — once daily
  Arms: Arm 1; Arm 2
Drug: matching placebo — once daily
  Arms: Arm 3; Arm 4

SUMMARY:
A multicentre, randomised, double-blind,4-stages phase III study enrolled 414 patients with chronic, previously treated ITP. Dosage could be adjusted (2.5~.75 mg/day) to maintain platelet counts 50~250×109/L

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of ITP ≥6 months;Platelets <30×109/L.
2. No evidence of other causes of thrombocytopenia.
3. Subjects who are refractory or have relapsed after at least one prior ITP therapy.
4. Previous therapy for ITP including rescue must have been completed at least 2 weeks prior to randomization.
5. Subjects treated with maintenance immunosuppressive therapy must be receiving a dose that has been stable for at least 1 month.
6. PT result no exceed normal by more than ±3s,APTT result no exceed normal by more than ±10s.
7. Signed informed consent.

Exclusion Criteria:

1. Patients with any prior history of arterial or venous thrombosis，or diagnosis as Thrombophilia.
2. Subjects diagnosed with tumor.
3. Have pre-existing cardiac disease within the last 3 months.No arrhythmia known to increase the risk of thrombolic events (e.g. atrial fibrillation), or patients with a Corrected QT interval (QTc) >450msec or QTc >480 for patients with a Bundle Branch Block.
4. Female subjects who are nursing or pregnant at screening or pre-dose on baseline.
5. Subjects who have previously received eltrombopag or any other thrombopoietin receptor agonist within 30 days .
6. Subject has consumed aspirin, aspirin-containing compounds, salicylates, anticoagulants, quinine or non-steroidal anti-inflammatories (NSAIDs) for >3 consecutive days within 2 weeks of the study start and until the end of the study.
7. Any laboratory or clinical evidence for HIV infection.Any clinical history for hepatitis C infection; chronic hepatitis B infection; or any evidence for active hepatitis at the time of subject screening.
8. ALT> 1.5 x upper limit of normal (ULN), AST> 3 x upper limit of normal (ULN)) DBLI> 1.2 x upper limit of normal (ULN),Scr> 1.2 x upper limit of normal (ULN)
9. The subject has participated in other clinical trial within the 3 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with a platelet count ≥50×109/L after Day 57. | Baseline to Week 8

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Union Hospital Tongji Medical College Huazhong University of Science and technology, Wuhan, Hubei
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Hospital of Blood Diseases, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Mei H, Liu X, Li Y, Zhou H, Feng Y, Gao G, Cheng P, Huang R, Yang L, Hu J, Hou M, Yao Y, Liu L, Wang Y, Wu D, Zhang L, Zheng C, Shen X, Hu Q, Liu J, Jin J, Luo J, Zeng Y, Gao S, Zhang X, Zhou X, Shi Q, Xia R, Xie X, Jiang Z, Gao L, Bai Y, Li Y, Xiong J, Li R, Zou J, Niu T, Yang R, Hu Y. Dose tapering to withdrawal stage and long-term efficacy and safety of hetrombopag for the treatment of immune thrombocytopenia: Results from an open-label extension study. J Thromb Haemost. 2022 Mar;20(3):716-728. doi: 10.1111/jth.15602. Epub 2021 Dec 15. PMID 34821020
- [Derived] Mei H, Liu X, Li Y, Zhou H, Feng Y, Gao G, Cheng P, Huang R, Yang L, Hu J, Hou M, Yao Y, Liu L, Wang Y, Wu D, Zhang L, Zheng C, Shen X, Hu Q, Liu J, Jin J, Luo J, Zeng Y, Gao S, Zhang X, Zhou X, Shi Q, Xia R, Xie X, Jiang Z, Gao L, Bai Y, Li Y, Xiong J, Li R, Zou J, Niu T, Yang R, Hu Y. A multicenter, randomized phase III trial of hetrombopag: a novel thrombopoietin receptor agonist for the treatment of immune thrombocytopenia. J Hematol Oncol. 2021 Feb 25;14(1):37. doi: 10.1186/s13045-021-01047-9. PMID 33632264